CLINICAL TRIAL: NCT03590093
Title: Enamel Matrix Derivatives on Systemic Inflammation After Periodontal Surgical Therapy
Brief Title: Amelogenins and Systemic Inflammation After Periodontal Surgical Therapy
Acronym: PERIOEMD-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, Clinical Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3649/13A
Record Dates: First submitted 2018-07-04; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The examiner were not aware of group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontal Surgery with EMD (Experimental): A surgical periodontal flap was elevated, degranulation of inflammatory tissues and dental debridement was performed. After carefully cleaning root dental surfaces, EMD was placed inside the infrabony periodontal defect. Suture were placed to maintain wound stability.
  Interventions: Procedure: Periodontal surgery; Procedure: EMD application
- Periodontal Surgery (Active Comparator): A surgical periodontal flap was elevated, degranulation of inflammatory tissues and dental debridement was performed. Suture were placed to maintain wound stability.
  Interventions: Procedure: Periodontal surgery

INTERVENTIONS:
Procedure: Periodontal surgery — After local anesthesia injection an intrasulcular flap is designed according to minimally invasive techniques. After flap elevation, careful removal of granulation tissues from the periodontal defects is performed. Scaling and root planing of the involved dental roots is ensured and finally suture is placed.
  Other Names: Open Flap Debridement
Procedure: EMD application — Application of Pref-Gel for 2 minutes and then the application on Enamel Matrix Derivatives on the surgically exposed root surface
  Other Names: Amelogenins application
  Arms: Periodontal Surgery with EMD

SUMMARY:
The aim of this study is to compare surgical treatment of periodontal infrabony defects with and without the adjunct of an enemal matrix derivative (EMD) in terms of acute-phase responses, in systemic healthy patients.

ELIGIBILITY:
Inclusion Criteria:

* Good health
* No previous periodontal surgical treatment
* Indication for periodontal surgery (intrabony defects to be at least 4 mm deep)
* Ability to understand the study procedures and comply with them through the length of the study

Exclusion Criteria:

* Pregnancy, breast feeding or taking oral contraceptive (all non-drug contraceptives will be allowed)
* The need for antibiotic therapy to undergo periodontal therapy
* Chronic infections
* Systemic diseases
* Patients who report current smoking over 20 cigarettes per day or pipe or cigar

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change of C Reactive Protein (CRP) at 24 hour | Collected at Baseline and 24 hours in order to calculate the changes
  CRP analyzed though blood sampling. Unit of measure: mg/L

SECONDARY OUTCOMES:
Glucose | Analyzed at Baseline, 24 hours, 1 week and 6 months after treatment
  analyzed though blood sampling. Unit of measure: mg/dL
Cholesterol | Analyzed at Baseline, 24 hours, 1 week and 6 months after treatment
  analyzed though blood sampling. Unit of measure: mg/dL
Triglycerides | Analyzed at Baseline, 24 hours, 1 week and 6 months after treatment
  analyzed though blood sampling. Unit of measure: mg/dL
HDL Cholesterol | Analyzed at Baseline, 24 hours, 1 week and 6 months after treatment
  analyzed though blood sampling. Unit of measure: mg/dL
LDL Cholesterol | Analyzed at Baseline, 24 hours, 1 week and 6 months after treatment
  analyzed though blood sampling. Unit of measure: mg/dL
Fibrinogen | Analyzed at Baseline, 24 hours, 1 week and 6 months after treatment
  analyzed though blood sampling. Unit of measure: mg/dL
D-Dimer | Analyzed at Baseline, 24 hours, 1 week and 6 months after treatment
  analyzed though blood sampling. Unit of measure: mg/L
Cystatin C | Analyzed at Baseline, 24 hours, 1 week and 6 months after treatment
  analyzed though blood sampling. Unit of measure: mg/L
C Reactive Protein (CRP) | Analyzed at Baseline, 24 hours, 1 week and 6 months after treatment
  CRP analyzed though blood sampling. Unit of measure: mg/L
Clinical attachment level (CAL) at deepest site | Measured at Baseline and 6 months after treatment
  Changes in CAL , measured orally through clinical examination. Unit of measure: mm
Pocket probing depth (PPD) at deepest site | Measured at Baseline and 6 months after treatment
  Changes in PPD , measured orally through clinical examination. Unit of measure: mm
Recession of the gingival margin (REC) | Measured at Baseline and 6 months after treatment
  Changes in REC, measured orally through clinical examination. Unit of measure: mm

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Graziani F, Peric M, Marhl U, Petrini M, Bettini L, Tonetti M, Gennai S. Local application of enamel matrix derivative prevents acute systemic inflammation after periodontal regenerative surgery: A randomized controlled clinical trial. J Clin Periodontol. 2020 Jun;47(6):747-755. doi: 10.1111/jcpe.13270. Epub 2020 Mar 12. PMID 32163634